CLINICAL TRIAL: NCT04030182
Title: Vitamin D Deficit in Women With Uterine Fibroids
Status: Completed | Type: Observational
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Luis Esteban González Varela, Gynecology Specialist, Adscript to the Gynecology Service in Regional General Hospital #45, Instituto Mexicano del Seguro Social
Other Study IDs: VIDANFI
Record Dates: First submitted 2019-07-02; First posted 2019-07-23 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Leiomyoma; Vitamin D Deficiency; Fibroid Uterus
MeSH Terms: conditions — Leiomyoma; Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — 3 ml of venous blood sample to determine levels of vitamin D
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Level of vitamin D: Level in blood sample of vitamin D for each patient
  Interventions: Diagnostic Test: Level of Vitamin D

INTERVENTIONS:
Diagnostic Test: Level of Vitamin D — 3 ml of venous blood will be taken to determine the level of vitamin D

SUMMARY:
Determinate the level of vitamin D in blood, and evaluate the prevalence of deficit and insufficiency among patients with diagnosis of uterine fibroids

DETAILED DESCRIPTION:
A cross-sectional prevalence study will be carried out, taking patients with a diagnosis of uterine fibroid in two hospitals; blood level of vitamin D will be taken to determine the proportion of patients with deficit and insufficiency; In addition, the number, size and type (according to the PALM-COEN classification) of the uterine fibroids in each patient will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Diagnosis of uterine fibroid

Exclusion Criteria:

* Female with diagnosis of uterine fibroid under treatment with exogenous vitamine D

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women with uterus and diagnosis of Uterine Leyomioma
Study Population: All female patients diagnosed with uterine myomatosis who come for consultation, if they agree to be part of protocol, an informed consent will be given and a 3 ml sample of venous blood will be taken.
  The present study will be performed in two Hospitals:
  "Centro Médico Nacional de Occidente" (CMNO) "Hospital General Regional No. 45" (HGR 45) Both hospital established in the city of Guadalajara, Jalisco, Mexico.
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-10-09 (Actual); Study Completion 2021-10-09 (Actual)

PRIMARY OUTCOMES:
appointment for intervention | 15 minutes
  All patients diagnosed with uterine fibroids who come for consultation, will be explained the protocol and if they agree to be part of it, an informed consent will be given and a 3 ml sample of venous blood will be taken.
  The sample will be analize in a COBAS 6000 ANALYZER SERIES model c501 (by ROCHE) and the reference levels will be:
  1-25 ng/mL - DEFICIT 25 - 30 ng/mL - INSUFFICIENCY > 30 ng/mL - Normal
  For this study, the qualitative variables will be expressed as frequencies and percentages (%); the quantitative variables will be expressed in means ± standard deviation. The prevalence of vitamin D deficiency at baseline will be calculated using the formula (total cases observed with vitamin D deficiency / total of patients included) X 100.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Esteban Gonzalez Varela, PhD, Principal Investigator — Instituto Mexicano del Seguro Social
Locations (2):
- Mexico (2):
  - Centro Médico Nacional de Occidente, Hospital de Gineco-Obstetricia, Guadalajara, Jalisco
  - Hospital General Regional No. 45, Guadalajara, Jalisco

IPD SHARING:
Plan to Share IPD: No
because is an internal study in the hospital, and the committe doesn´s accept share any information

REFERENCES:
- [Background] Blauer M, Rovio PH, Ylikomi T, Heinonen PK. Vitamin D inhibits myometrial and leiomyoma cell proliferation in vitro. Fertil Steril. 2009 May;91(5):1919-25. doi: 10.1016/j.fertnstert.2008.02.136. Epub 2008 Apr 18. PMID 18423458
- [Background] Pavone D, Clemenza S, Sorbi F, Fambrini M, Petraglia F. Epidemiology and Risk Factors of Uterine Fibroids. Best Pract Res Clin Obstet Gynaecol. 2018 Jan;46:3-11. doi: 10.1016/j.bpobgyn.2017.09.004. Epub 2017 Oct 1. PMID 29054502
- [Background] Lukes AS, Soper D, Harrington A, Sniukiene V, Mo Y, Gillard P, Shulman L. Health-Related Quality of Life With Ulipristal Acetate for Treatment of Uterine Leiomyomas: A Randomized Controlled Trial. Obstet Gynecol. 2019 May;133(5):869-878. doi: 10.1097/AOG.0000000000003211. PMID 30969201
- [Result] Holick MF, Binkley NC, Bischoff-Ferrari HA, Gordon CM, Hanley DA, Heaney RP, Murad MH, Weaver CM; Endocrine Society. Evaluation, treatment, and prevention of vitamin D deficiency: an Endocrine Society clinical practice guideline. J Clin Endocrinol Metab. 2011 Jul;96(7):1911-30. doi: 10.1210/jc.2011-0385. Epub 2011 Jun 6. PMID 21646368
- [Result] Cashman KD, Sheehy T, O'Neill CM. Is vitamin D deficiency a public health concern for low middle income countries? A systematic literature review. Eur J Nutr. 2019 Feb;58(1):433-453. doi: 10.1007/s00394-018-1607-3. Epub 2018 Jan 17. PMID 29344677
- [Result] Atkinson SA. [The new dietary reference intakes from the Institute of Medicine for calcium and vitamin D]. Perspect Infirm. 2011 Sep-Oct;8(5):5. No abstract available. French. PMID 21939083
- [Result] Halder S, Al-Hendy A. Hypovitaminosis D and high serum transforming growth factor beta-3: important biomarkers for uterine fibroids risk. Fertil Steril. 2016 Dec;106(7):1648-1649. doi: 10.1016/j.fertnstert.2016.09.048. Epub 2016 Oct 25. No abstract available. PMID 27793369
- [Result] Jukic AM, Steiner AZ, Baird DD. Lower plasma 25-hydroxyvitamin D is associated with irregular menstrual cycles in a cross-sectional study. Reprod Biol Endocrinol. 2015 Mar 11;13:20. doi: 10.1186/s12958-015-0012-5. PMID 25879830
- [Result] Protic O, Toti P, Islam MS, Occhini R, Giannubilo SR, Catherino WH, Cinti S, Petraglia F, Ciavattini A, Castellucci M, Hinz B, Ciarmela P. Possible involvement of inflammatory/reparative processes in the development of uterine fibroids. Cell Tissue Res. 2016 May;364(2):415-27. doi: 10.1007/s00441-015-2324-3. Epub 2015 Nov 27. PMID 26613601
- [Result] Skowronska P, Pastuszek E, Kuczynski W, Jaszczol M, Kuc P, Jakiel G, Woclawek-Potocka I, Lukaszuk K. The role of vitamin D in reproductive dysfunction in women - a systematic review. Ann Agric Environ Med. 2016 Dec 23;23(4):671-676. doi: 10.5604/12321966.1226865. PMID 28030942
- [Result] Holick MF. Vitamin D: A millenium perspective. J Cell Biochem. 2003 Feb 1;88(2):296-307. doi: 10.1002/jcb.10338. PMID 12520530
- [Result] Ali, M. et al. Vitamin D synergizes the antiproliferative, apoptotic, antifibrotic and anti-inflammatory effects of ulipristal acetate against human uterine fibroids Fertility and Sterility, Volume 108, Issue 3, e66
- [Result] Hartmann KE, Fonnesbeck C, Surawicz T, Krishnaswami S, Andrews JC, Wilson JE, Velez-Edwards D, Kugley S, Sathe NA. Management of Uterine Fibroids [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2017 Dec. Report No.: 17(18)-EHC028-EF. Available from http://www.ncbi.nlm.nih.gov/books/NBK537742/ PMID 30789683
- [Result] Munro MG, Critchley HO, Broder MS, Fraser IS; FIGO Working Group on Menstrual Disorders. FIGO classification system (PALM-COEIN) for causes of abnormal uterine bleeding in nongravid women of reproductive age. Int J Gynaecol Obstet. 2011 Apr;113(1):3-13. doi: 10.1016/j.ijgo.2010.11.011. Epub 2011 Feb 22. PMID 21345435
- [Result] Styer AK, Rueda BR. The Epidemiology and Genetics of Uterine Leiomyoma. Best Pract Res Clin Obstet Gynaecol. 2016 Jul;34:3-12. doi: 10.1016/j.bpobgyn.2015.11.018. Epub 2015 Dec 2. PMID 26725703
- [Result] Dubuisson J. The current place of mini-invasive surgery in uterine leiomyoma management. J Gynecol Obstet Hum Reprod. 2019 Feb;48(2):77-81. doi: 10.1016/j.jogoh.2018.10.004. Epub 2018 Oct 12. PMID 30316905
- [Result] Borah BJ, Nicholson WK, Bradley L, Stewart EA. The impact of uterine leiomyomas: a national survey of affected women. Am J Obstet Gynecol. 2013 Oct;209(4):319.e1-319.e20. doi: 10.1016/j.ajog.2013.07.017. Epub 2013 Jul 24. PMID 23891629